



## Study Protocol

Study Title: Portal Vein Flow Variability to Quantify Right-Sided Hemodynamic Congestion: A Proof-

Of-Concept study

Study Acronym: PORTAL Phase of Development: N/A

**Protocol Number: 3** 

Protocol Version and Date: Version 3.0, May 30th, 2022

**EudraCT Registry Number: N/A** ClinicTrials.gov Registry Number: Investigational product: None

**Sponsor:** UZ Brussel

Coordinating/Principal Investigator: Prof. Dr. Frederik Verbrugge

The information contained in this document is the property of the Sponsor/Coordinating Investigator and may not be reproduced, published or disclosed to others without written authorization of the Sponsor/Coordinating Investigator.

#### PROTOCOL SIGNATURE PAGE

Protocol Version and date: Version 3.0, May 30th, 2022

Protocol Title: Portal Vein Flow Variability to Quantify Right-Sided Hemodynamic Congestion: A

Proof-Of-Concept study

**Sponsor:** UZ Brussel

Principal Investigator: Prof. Dr. Frederik Verbrugge

#### I agree:

- to assume responsibility for the proper conduct of this study
- to conduct the study in compliance with this protocol and any future amendments
- not to implement any deviations from or changes to the protocol without prior review and written approval from the Ethics Committee, except where necessary to eliminate an immediate hazard to the subjects, or for administrative aspects of the study (where permitted by all applicable regulatory requirements)
- that I am thoroughly familiar with the appropriate use of the investigational drug, as described in this protocol
- to ensure that all persons assisting me with the study are adequately informed about the investigational drug and their study-related duties and functions as described in the protocol
- that I am aware of and will comply with the current good clinical practice (GCP) guidelines and ethical principles outlined in the Declaration of Helsinki

to conduct the study in accordance with all applicable laws and regulations

Date: 30/05/2022 Printed name: Frederik Verbrugge Signature

Version 3.0, 30/05/2022

1/4| Page





#### Study Protocol

# Portal Vein Flow Variability to Quantify Right-Sided Hemodynamic Congestion (PORTAL):

### A Proof-Of-Concept study

Simon Vanhentenrijk M.D. Pharm.D. & Frederik H. Verbrugge M.D. Ph.D.

#### 1. Study design

- Prospective
- Interventional
- Single centre (UZ Brussel)
- Proof-of-concept

#### 2. Purpose & rationale

Right ventricular hemodynamic congestion or elevated central venous pressure (CVP) is an independent predictor of morbidity and mortality in heart failure (1). Persistent elevations of right atrial pressure (RAP) cause upstream venous congestion in the abdominal compartment, which leads to organ dysfunction in liver and kidney function, with effects on the lungs as well (2), (3). According to contemporary echocardiography guidelines, non-invasive assessment of RAP is performed by measuring inferior vena cava (IVC) size and respiratory variation (i.e., collapsibility) (4). However, assumptions that are not always valid (especially in critically ill patients) hamper the use of this technique and misinterpretation due to 'pseudo-collapse' could lead to erroneous interpretation.





Portal vein Doppler flow patterns may be a simple and attractive tool to aid in the evaluation of RAP/CVP and predicts acute kidney injury after cardiac surgery (5). The aim of this proof-of-concept study is to assess the feasibility of portal vein Doppler flow to quantify RAP/CVP in a population of consecutive patients with advanced heart failure undergoing invasive right heart catheterization.

#### 3. Objective

To evaluate the accuracy of the portal vein pulsatility index (PVPI=Vmax-Vmin)/Vmax) to quantify invasively measured right-sided venous pressures.

#### 4. Study population

#### a. Inclusion criteria

- At least 18 y/o and able to provide informed consent
- Consecutive patients scheduled for right heart catheterisation by a dedicated heart failure specialist at the Centre of Cardiovascular Diseases (University Hospital Brussels, Jette, Belgium)

#### b. Exclusion criteria

- Major anatomical variations of the portal veins (agenesis of left and right portal vein) and/or arterio-portal vein fistula
- Patients with Child-Pugh B or C liver cirrhosis or liver transplant
- Body Mass Index < 20 kg/m²</li>

#### 5. Intervention

All patients will undergo right heart catheterisation for clinical reasons. As part of the hemodynamic assessment, RAP and CVP assessed at the level of the intrathoracic and intra-abdominal IVC as well as the vena Hepatica is measured. In addition, the hepatic venous wedge pressure (HVWP) is measured.

PVPI is simultaneously obtained using point-of-care ultrasound by placing the transducer at the right hypochondrium/right lateral region of the corpus. Portal vein flow velocity is obtained by using pulsed





wave Doppler measurements of the left portal vein. In addition, a non-invasive measuring device to assess the mechanical energy of the heart by registering its vibrations (i.e., Kinocardiography, HeartKinetics, Waterloo, Belgium) is put on the participant with sticky-gel electrodes. A 90-second measurement is done once the patient is in the supine position. The same measurement is performed simultaneously by a smartphone application with the smartphone placed centrally on the participant's chest.

To minimize interobserver variability, the same sonographic equipment will be used by the same, independent researcher. Measurements are obtained in supine position at the end of the respiratory cycle (end-expiratory). In order to correlate the study outcome with clinical situations, demographic characteristics of the participants are collected.

#### 6. Safety precautions

There are no known risks except for those of the clinically indicated right heart catheterisation. Echocardiography can cause local discomfort and in rare occasions contusion from local pressure. The Kinocardiography device is completely non-invasive as well, although theoretically, there might be some skin irritation due to its attachment with sticky-gel electrodes.

#### 7. Statistical analysis

#### a. Main statistical analysis

The correlation between PVPI and RAP, CVP and HVWP will be assessed by classic regression and Bland-Altman plots. A regression formula for RAP will be constructed based on PVPI and age, gender, height and weight if the latter are contributory.

#### 8. References

- 1. Binanay C, Califf RM, Hasselblad V, O'Connor CM, Shah MR, Sopko G, et al. Evaluation study of congestive heart failure and pulmonary artery catheterization effectiveness: the ESCAPE trial. Jama. 2005;294(13):1625-33.
- 2. Verbrugge FH, Guazzi M, Testani JM, Borlaug BA. Altered Hemodynamics and End-Organ Damage in Heart Failure: Impact on the Lung and Kidney. Circulation. 2020;142(10):998-1012.
- 3. Verbrugge FH, Dupont M, Steels P, Grieten L, Malbrain M, Tang WH, et al. Abdominal contributions to cardiorenal dysfunction in congestive heart failure. J Am Coll Cardiol. 2013;62(6):485-95.





- 4. Porter T, Shillcutt S, Adams M, Desjardins G, Glas K, Olson J, Troughton R, et al. Guidelines for the use of echocardiography as a monitor for therapeutic intervention in adults: a report from the American Society of Echocardiography. J Am Soc Echocardiogr. 2015 Jan;28(1):40-56.
- 5. Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, et al. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020;12(1):16.